CLINICAL TRIAL: NCT05711992
Title: Rare Embryonal Tumors of the Central Nervous System: International Registry
Status: Recruiting | Type: Observational
Sponsor: Immune Oncology Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IMMONC0005
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Embryonal Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Central nervous system (CNS) tumors are the most common solid malignancies among children. Although some types of CNS tumors like medulloblastomas and low-grade gliomas are widespread and well-studied, there is a huge number of rare diseases that need further research. This international registry aims to establish a large multicenter database of pediatric and young adult patients with rare embryonal tumors of the central nervous system and describe the clinical presentations, diagnostics, treatment regimens, and outcomes. Embryonal tumors with multilayered rosettes (ETMR), FOXR2-activated CNS neuroblastoma, cribriform neuroepithelial tumor, and CNS tumor with BCOR internal tandem duplication are extremely rare embryonal tumors some of which were first described in the last edition of the World Health Organization (WHO) Classification of Tumors of the Central Nervous System. Objectives of the registry are 1) to evaluate prognostic factors, 2) to identify diagnostic and treatment gaps, 3) to investigate the characteristics and outcome of the disease with different treatment regimens, and 4) to generate data-based prospective diagnostic and treatment recommendations.

DETAILED DESCRIPTION:
CNS tumors are the most common solid malignancies and the leading cause of children's cancer-related mortality. Embryonal tumors account for approximately 20-25% of all primary CNS tumors in children. Although medulloblastomas are the most commonly diagnosed malignant brain tumors, other embryonal tumors are relatively rare. Several studies of rare embryonal tumors have been published, but the number of included patients is generally small. Diagnosis of different subtypes of rare embryonal tumors can be extremely challenging. Because of limited data, there are no standard treatment recommendations for patients with rare embryonal tumors.

Embryonal tumors with multilayered rosettes (ETMR), FOXR2-activated CNS neuroblastoma, cribriform neuroepithelial tumor, CNS tumor with BCOR internal tandem duplication, and embryonal tumors not otherwise specified/not elsewhere classified (NOS/NEC) are extremely rare. Moreover, FOXR2-activated CNS neuroblastoma, cribriform neuroepithelial tumor, and CNS tumor with BCOR internal tandem duplication were first described in the fifth edition of the WHO Classification of Tumors of the Central Nervous System, published in 2021. Because of the rarity of these tumors, randomized controlled clinical trials are extremely complicated to conduct. Considering the lack of studies from low- and middle-income countries (LMICs) it is not excluded that cases of rare embryonal tumors are more common than have been described in the literature. Hence, evidence can be generated through registry studies.

This is a multicenter international retrospective and prospective registry to collect and analyze data from pediatric and young adult patients diagnosed with rare CNS embryonal tumors. Patients will be recruited directly by participating centers and national study groups. Participating centers will collect and verify the informed consent of all prospective patients enrolled at their centers.

Patients diagnosed with rare embryonal tumors of the CNS (ETMR, FOXR2-activated CNS neuroblastoma, cribriform neuroepithelial tumor, CNS tumor with BCOR internal tandem duplication, embryonal tumors NOS/NEC) since 01.01.2010 will be included. ETMR has been included in the WHO classification of CNS tumors since 2016 and encompasses three morphologically distinct embryonal tumors (Embryonal tumor with abundant neuropil and true rosettes (ETANTR), ependymoblastoma (EBL) and medulloepithelioma (MEPL)) that were previously classified as CNS primitive neuroectodermal tumors (CNS-PNETs). These histological subtypes should also be included in the study. Considering the lack of molecular genetic tests done among retrospective cases, the investigators will also include all patients diagnosed with neuroblastoma and ganglioneuroblastoma.

The following data will be collected through questionnaires:

1. Patient characteristics
2. Characteristics of rare CNS embryonal tumors
3. Details of the diagnosis and treatment
4. Complications and late effects of treatment
5. Outcomes
6. Follow-up information

Quality control and data management will be conducted by the Immune Oncology Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rare embryonal tumors of CNS since 01.01.2010:

  * ETMR (including embryonal tumor with abundant neuropil and true rosettes (ETANTR), ependymoblastoma (EBL) and medulloepithelioma (MEPL) which were previously classified as CNS-PNETs)
  * FOXR2-activated CNS neuroblastoma
  * cribriform neuroepithelial tumor
  * CNS tumor with BCOR internal tandem duplication
  * all patients diagnosed with neuroblastoma and ganglioneuroblastoma with no molecular genetic tests available
* Patients ≤ 25 years of age
* Signed informed consent form for prospective patients ≥ 18 years of age
* Signed parental permission and child assent forms for prospective patients < 18 years of age

Exclusion Criteria:

• CNS metastases of extracranial embryonal tumors

Ages: 1 Day to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients diagnosed with rare embryonal tumors
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2033-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years
5-year overall survival | 5 years

SECONDARY OUTCOMES:
Complete remission rate | 5 years
3-year event-free survival | 3 years
5-year event-free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Julieta Hoveyan, MD, Principal Investigator — Immune Oncology Research Institute, Yerevan, Armenia; Ruzanna Papyan, MD, Principal Investigator — Immune Oncology Research Institute, Yerevan, Armenia; Gevorg Tamamyan, MD, PhD, DSc, Study Director — Immune Oncology Research Institute, Yerevan, Armenia
Locations (11):
- Hematology Center named after prof. R. Yeolyan, Yerevan, Armenia
- Children's Hospital of Eastern Ontario (CHEO), Ottawa, Canada
- Semmelweis University, Budapest, Hungary
- National Cancer Institute, All India Institutes of Medical Sciences, New Delhi, India
- Oncology Department of Golestan hospital, Tehran, Iran
- IRCCS Istituto Ospedale Pediatrico Bambino Gesù, Rome, Italy
- Mexico (2):
  - Hospital Civil de Guadalajara "Dr. Juan I. Menchaca", Guadalajara
  - Centro Médico ABC, Mexico City
- Peru (2):
  - Hospital Nacional Alberto Sabogal Sologuren - EsSalud, Bellavista
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
- China Medical University Children's Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided